CLINICAL TRIAL: NCT00115921
Title: Evaluation of Home-Based Management of Fever in Urban Ugandan Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Makerere University (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCRVG40
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria; Anemia
Keywords: Home-based care; Malaria; Africa
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Provision of antimalarial treatment at home

SUMMARY:
The purpose of this study is to see if providing effective antimalarial treatment at home for parents/guardians to treat their children for malaria will lead to an improved health outcome compared to conventional healthcare.

DETAILED DESCRIPTION:
Population: Representative sample of Ugandan children aged 1 to 5 years from 400 households (approximately 540 children).

Clinical Site: The study will be conducted in the Mulago III parish community of Kampala, Uganda.

Study Duration: 13 months

Study Intervention: *Pilot period: After enrollment, households will participate in a one month pilot period to test the household pictorial diaries. At the end of the pilot period, households will be randomized to participation in the home-based management of fever (HBMF) arm or standard care arm for the remainder of the study (12 months). *HBMF arm: Households randomized to the HBMF group will be provided with pre-packaged coartemether to keep at home. Primary caregivers will be instructed to treat children participating in the study empirically with coartemether at home when the child develops fever. Study personnel will distribute drugs and educate the caregivers about administration of drugs, recognition of danger signs of fever/malaria, and when to seek additional care. *Standard care: Households randomized to the standard care arm will be asked to continue their current behaviour and to manage fever in their children as they would normally.

Measurements: Household diaries and monthly visits. Primary caregivers will be asked to keep a diary regarding the health of study participants for the duration of the study (13 months). Information on illnesses, treatments given, visits to health care facilities, and health care expenditures will be collected. Study personnel will visit the households monthly to collect completed diaries. At each visit, questionnaires will be administered to gather additional data on the health of the participants and treatment seeking behaviour.

Clinical and laboratory evaluations: Temperature, height, weight, mid-upper arm circumference, spleen size, haemoglobin, and thick blood smear will be assessed at enrollment, and at the beginning and end of the intervention period.

Study Objectives: 1. To measure the impact of home-based management of fever with coartemether on malaria-related morbidity compared to the current standard of care in the community.

2. To measure the impact of home-based management of fever with coartemether on economic measures compared to the current standard of care in the community.

Primary outcome: Treatment incidence density (treatments per time at risk) for each treatment arm

Secondary clinical outcomes: 1) mean days of fever; 2) incidence of febrile episodes; 3) mean haemoglobin at study end; 4) change in mean haemoglobin; 5) prevalence of splenomegaly; 6) prevalence of parasitaemia; 7) incidence of visits to health care facilities, and hospitalizations; 8) mortality rate; 9) anthropometric measurements; 10) proportion of "appropriate" treatments; 11) proportion of delayed treatments; 12) treatment incidence density of treatments given at >50% and at full dose

Economic outcomes: 1) household cost/febrile episode; 2) household costs for treatment of febrile episode/month; 3) provider cost/child for delivery of HBMF; 4) estimated provider facility cost/patient for uncomplicated fever, and for severe disease; 5) total net cost/child/year; 6) net cost/additional child appropriately treated; 7) net cost/day of fever averted

ELIGIBILITY:
Inclusion Criteria:

* Age 1 - 5 years
* Agreement of parents or guardians to provide informed consent
* Live in Mulago III Parish

Exclusion Criteria:

* History of any known serious chronic disease requiring frequent medical care (e.g. AIDS, sickle cell disease, malignancy)
* Intention to move from Kampala during the 13 month follow-up period
* History of serious side effects to study medications
* Weight < 10 kg
* Severe malnutrition defined as a weight-for-height or height-for-age Z-score < - 3

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 540
Dates: Start 2005-07; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measurement will be treatment incidence density (antimalarial treatments received per time at risk) for each study arm.

SECONDARY OUTCOMES:
Mean days of fever per participant
Incidence of febrile episodes
Mean haemoglobin at study end
Change in mean haemoglobin between the start and end of the intervention
Incidence of visits to health care facilities (drug shops, clinics, pharmacies, hospitals) and hospitalizations per participant
Mortality rate
Economic outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Sarah G Staedke, MD, Principal Investigator — University of California, San Francisco; Christopher JM Whitty, FRCP, Principal Investigator — London School of Hygiene and Tropical Medicine

REFERENCES:
- [Derived] Staedke SG, Mwebaza N, Kamya MR, Clark TD, Dorsey G, Rosenthal PJ, Whitty CJ. Home management of malaria with artemether-lumefantrine compared with standard care in urban Ugandan children: a randomised controlled trial. Lancet. 2009 May 9;373(9675):1623-31. doi: 10.1016/S0140-6736(09)60328-7. Epub 2009 Apr 9. PMID 19362361